CLINICAL TRIAL: NCT05705804
Title: Effects of Pitavastatin or Combination of Pitavastatin and Ezetimibe on Glucose Metabolism Compared to AtoRvastatin in atheroscLerotic Cardiovascular Disease Patients With Metabolic Syndrome: The EZ-PEARL Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1325
Record Dates: First submitted 2023-01-18; First posted 2023-01-31 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Dyslipidemias; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group P (Experimental): Pitavastatin 4mg group
  Interventions: Drug: Pitavastatin
- Group PE (Experimental): Pitavastatin 4 mg Ezetimibe 10 mg combined administration group
  Interventions: Drug: Pitavastatin plus Ezetemibe
- Group A (Active Comparator): Atorvastatin 40 mg administration group
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4 mg will be given.
  Arms: Group P
Drug: Pitavastatin plus Ezetemibe — Pitvastatin 4 mg plus ezetemibe 10 mg will be given.
  Arms: Group PE
Drug: Atorvastatin — Atorvastatin 40 mg will be given.
  Arms: Group A

SUMMARY:
The purpose of this study was to investigate the effect of pitavastatin or pitavastatin and ezetimibe combination therapy on glucose metabolism compared to atorvastatin in patients with atherosclerotic cardiovascular disease with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia
2. Patient with diagnosis of clinical atherosclerotic cardiovascular disease (acute coronary syndrome, history of myocardial infarction, stable or unstable angina, history of coronary artery reperfusion, stroke or transient stroke, history of peripheral arterial disease or peripheral arterial reperfusion)
3. Patients with metabolic syndrome but without diabetes

Exclusion Criteria:

1. Diagnosis of clinical atherosclerotic cardiovascular disease within 1 year
2. Acute liver disease or persistent unexplained serum AST or ALT three times the upper limit of normal
3. Allergy or hypersensitivity to statins or ezetimibe
4. Solid organ transplant recipients
5. History of side effects requiring discontinuation of statin administration
6. Pregnant women, potentially pregnant or lactating women
7. Life expectancy less than 3 years
8. If it is judged that follow-up for more than 1 year is not possible
9. If the patient is unable to understand or read the consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change form baseline homeostatic model assessment for insulin resistance (HOMA-IR) at 24 weeks | At 24 weeks
  Changes of homeostatic model assessment for insulin resistance (HOMA-IR) form baseline to 24 weeks will be compared among the three groups.

SECONDARY OUTCOMES:
Proportion of fasting glucose ≥100 mg/dL | At 24 weeks
Proportion of HbA1C ≥6.5% | At 24 weeks
Proportion of new-onset diabetes mellitus | At 24 weeks
Changes of HOMA-β at 24 weeks | At 24 weeks
Changes of fasting glucose at 24 weeks | At 24 weeks
Changes of insulin at 24 weeks | At 24 weeks
Changes of HbA1c at 24 weeks | At 24 weeks
Changes of triglyceride at 24 weeks | At 24 weeks
LDL-cholesterol change at 24 weeks | At 24 weeks
HDL-cholesterol change at 24 weeks | At 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, Principal Investigator — Severance Cardiovascular Hospital, YONSEI UNIVERSITY COLLEGE OF MEDICINE
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No